CLINICAL TRIAL: NCT05485584
Title: An International, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel, Phase II Pilot Study to Evaluate the Efficacy and Safety of Recombinant Super-compound Interferon (rSIFN-co) Among Healthy Subjects in Close Contact With Confirmed COVID-19 Case(s) and Subjects With Mild or Asymptomatic COVID-19
Brief Title: rSIFN-co Among Healthy Subjects and Subjects With Mild or Asymptomatic COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Huiyang Life Science and Technology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SHL-rSIFN-002
Record Dates: First submitted 2022-06-16; First posted 2022-08-03 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-04

CONDITIONS: COVID-19; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy subjects(A1) (Experimental): Each nostril: 2 sprays/time; Pharynx: 4 sprays/time; Once daily
  Interventions: Drug: rSIFN-co Nasal Spray
- Healthy subjects(A2) (Placebo Comparator): Each nostril: 2 sprays/time; Pharynx: 4 sprays/time; Once daily
  Interventions: Drug: Placebo Nasal Spray
- COVID-19 subjects(B1) (Experimental): Each nostril: 2 sprays/time; Pharynx: 4 sprays/time; Twice daily
  Interventions: Drug: rSIFN-co Nasal Spray
- COVID-19 subjects(B2) (Placebo Comparator): Each nostril: 2 sprays/time; Pharynx: 4 sprays/time; Twice daily
  Interventions: Drug: Placebo Nasal Spray

INTERVENTIONS:
Drug: rSIFN-co Nasal Spray — 8 million IU (16 μg)/day; Once daily
  Other Names: rSIFN-co
  Arms: Healthy subjects(A1)
Drug: rSIFN-co Nasal Spray — 16 million IU (32 μg)/day; Twice daily
  Other Names: rSIFN-co
  Arms: COVID-19 subjects(B1)
Drug: Placebo Nasal Spray — Once daily
  Other Names: ingredients
  Arms: Healthy subjects(A2)
Drug: Placebo Nasal Spray — Twice daily
  Other Names: ingredients
  Arms: COVID-19 subjects(B2)

SUMMARY:
This is a phase II pilot, international, multicenter, randomized, double-blind, placebo-controlled study that aims to evaluate the safety and preliminary efficacy of rSIFN-co nasal spray in healthy subjects in close contact with confirmed COVID-19 case(s) as well as subjects with mild or asymptomatic COVID-19.

DETAILED DESCRIPTION:
Approximately 200 subjects are planned to be enrolled, including 100 healthy subjects and 100 COVID-19 subjects.

For the healthy subjects in close contact with confirmed COVID-19 case(s) (Group A), approximately 100 subjects will be randomized in a 1:1 ratio to receive placebo or rSIFN-co treatment in a double-blind fashion.

For the subjects with mild or asymptomatic COVID-19 (Group B), approximately 100 subjects will also be randomly assigned in a 1:1 ratio to receive institutional or local standard of care (SoC) plus placebo or SoC plus rSIFN-co in a double-blind fashion.

All subjects will receive the study product for 10 days; around 8 million IU (16 μg) or 16 million IU (32 μg) of rSIFN-co will be administered daily. The safety and efficacy parameters will be monitored throughout the study period. Subjects will be instructed to complete a diary to record daily administration of study product, SpO2 level, as well as the occurrence and severity of any clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 and ≤75 years of age at the time of informed consent.
2. Willing and able to provide written informed consent/assent for the trial.
3. Healthy subjects in close contact with confirmed COVID-19 case(s) or subjects with mild or asymptomatic COVID-19.

   a. Healthy subjects in close contact with confirmed COVID-19 case(s) i. With exposure to confirmed COVID-19 case(s) within 96 hours (refer to the definition of healthy subjects in close contact with confirmed COVID-19 case[s]), ii. Negative reverse transcriptase-polymerase chain reaction (RT-PCR) test for SARS-CoV-2 infection, with the sample collected at screening, iii. Have no previous confirmed COVID-19 diagnosis, iv. Without symptoms of respiratory infection, including fever, cough, fatigue, anorexia, shortness of breath, myalgias, sore throat, nasal congestion, headache, gastrointestinal symptoms, loss of smell (anosmia), loss of taste (ageusia), or other symptoms associated with COVID-19, AND v. With stable health status, as judged by the investigator and determined by physical examination, vital signs, medical history, and laboratory tests at screening.

   b. Subjects with mild or asymptomatic COVID-19 i. Meeting the criteria of mild or asymptomatic COVID-19,

   Note:
   * Asymptomatic or presymptomatic infection: Individuals who test positive for SARS-CoV-2 by virologic testing using a molecular diagnostic (e.g., PCR) or antigen test, but have no symptoms.
   * Mild disease: Individuals who have any of the various signs and symptoms of COVID-19 (e.g., fever, cough, sore throat, malaise, headache, muscle pain) and saturation of oxygen (SpO2) ≥90% on room air at sea level, without shortness of breath, dyspnea, or abnormal chest imaging.

   ii. Positive RT-PCR test for SARS-CoV-2 infection, with the sample collected at screening or within 72 hours prior to screening, AND iii. Without evidence of viral pneumonia or hypoxia.
4. Women of childbearing potential must have a negative pregnancy test result at screening.
5. Males and females who are fertile must adhere to contraception requirements for the duration of the study.
6. Non-participation in any other clinical trials during the study period.

Exclusion Criteria:

1. Subjects with any of the following conditions that would impair their ability to participate reliably in the trial, or those who may increase the risk to themselves or others by participating

   1. Clinically significant laboratory abnormalities (including a screening test of aspartate aminotransferase/alanine aminotransferase (AST/ALT) > 5 times the upper limit of normal [ULN] and/or estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73m2)
   2. Serious medical illnesses (including known history of major hematological, renal, cardiovascular, or hepatic abnormalities that are clinically significant)
   3. Psychological condition or social circumstances
2. Received an experimental medication within 1 month prior to screening or expect to receive such treatment during the study period.
3. With contraindication or hypersensitivity to the study product or any of its component.
4. Pregnant or lactating women.
5. Unwilling or unable to follow protocol requirements.
6. Any condition which in the investigator's opinion deems the potential participant an unsuitable candidate to receive the study product.
7. Received any interferons and any nasal/pharyngeal sprays within 7 days prior to screening.
8. Received COVID-19 vaccine within 14 days prior to screening
9. Had previous confirmed SARS-CoV-2 infection >96 hours prior to being screened for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Incidence of laboratory-confirmed SARS-CoV-2 infection in health subjects | Day1-Day28
  Incidence of laboratory-confirmed SARS-CoV-2 infection in health subjects over 28 days (Day 1 to Day 28) as assessed by RT-PCR
Percentage of subjects with disease progression | Day1-Day28
  Percentage of subjects with disease progression, defined as progression from asymptomatic/mild to moderate/severe in severity, over 28 days

SECONDARY OUTCOMES:
To assess the safety and tolerability profiles of rSIFN-co nasal spray, as assessed by treatment-emergent adverse events (TEAEs) | Day1-Day28
  TEAEs will be coded using the Medical Dictionary for Drug Regulatory Affairs (MedDRA®, version 24.1 or later) and presented as summary tabulations, including categorical information of interest such as severity, causal relationship to study medication, and action taken.
Percentage of subjects discontinuing from study product due to TEAE during the treatment period | Day1-Day10
  All AEs will be assessed by the Investigator using the CTCAE version 5.0.
Percentage of subjects who develop to moderate or severe COVID-19 (WHO definition) over 28 days | Day1-Day28
  For healthy subjects only
Incidence of COVID-19-related complications over 28 days | Day1-Day28
  For healthy subjects only
Time to clearance of SARS-CoV-2 | Day1-Day28
  For COVID-19 subjects only. It defined as 2 consecutive negative swabs (sampling interval ≥24 hours)
Percentage of subjects who require supplemental oxygen or mechanical ventilation | Day1-Day28
  For COVID-19 subjects only.
Percentage of subjects with clinical improvement | Day1-Day10
  For COVID-19 subjects only. It defined as a decrease of at least one point per the 11-point WHO clinical progression scale compared to baseline, on Days 5 and 10
Time to clinical improvement from the highest outcome scores per 11-point WHO clinical progression scale | Day1-Day28
  For COVID-19 subjects only.
Time to resolution of all symptoms present at baseline | Day1-Day28
  For COVID-19 subjects only.

CONTACTS AND LOCATIONS:
Overall Officials: GW WEI, Study Director — Sichuan Huiyang Life Science and Technology Corporation
Locations (2):
- Philippines (2):
  - GreenCity Medical Center, San Fernando City, Central Luzon
  - Medical Center Manila, Manila